CLINICAL TRIAL: NCT03510767
Title: A Phase I Study of TQ-B3525 on Tolerance and Pharmacokinetics
Brief Title: A Study of TQ-B3525 on Tolerance and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-I-01
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Relapsed or Refractory Lymphoma or Advanced Cancer
MeSH Terms: conditions — Recurrence; Lymphoma | interventions — TQ-B3525

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 (Experimental)
  Interventions: Drug: TQ-B3525

INTERVENTIONS:
Drug: TQ-B3525 — TQ-B3525 p.o. qd

SUMMARY:
To study the pharmacokinetic characteristics of TQ-B3525 in the human body, recommend a reasonable regimen for subsequent research.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory lymphoma or advanced solid tumor that diagnosed Pathologically or cytologically diagnosed
* ECOG PS≤1
* Adequate blood cell counts, kidney function and liver function
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Patients with immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or organ transplant history
* Hypertension (systolic BP ≥150 mmHg, diastolic BP ≥90 mmHg) still uncontrollable by one medication
* Hepatitis B virus patients with active replication (DNA> 500 cps / mL), hepatitis C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLT) | Baseline up to 28 days
  DLT: An adverse event occurring after initiation of TQ-B3525 that met any following criteria:
  1. >=Grade 3 of non-hematology toxicity
  2. Grade 4 hematology toxicity
Maximum Tolerated Dose (MTD) | Baseline up to 28 days
  MTD was defined as the highest dose level studied for which the incidence of first cycle DLT was < 33%.

CONTACTS AND LOCATIONS:
Overall Officials: Huaqing Wang, doctor, Study Chair — People's Hospital of Tianjin Tianjin,China,300121; Wenqi Jiang, doctor, Study Chair — Sun Yat-sen University Cancer Center,Guangzhou,Guangdong,China, 510060
Locations (1):
- People's Hospital of Tianjin, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided